CLINICAL TRIAL: NCT06629675
Title: Personalised Music Feedback to Optimise Adherence to the Walking Exercise Prescription During Pulmonary Rehabilitation for Individuals Living With Chronic Obstructive Pulmonary Disease
Brief Title: Make Every Step Count: Personalised Music Feedback to Walking for People Living With COPD
Acronym: MuSiC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University of Strathclyde (Other); University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0976
Record Dates: First submitted 2024-09-26; First posted 2024-10-08 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Chronic Obstructive Lung Disease; Chronic Obstructive Airway Disease
Keywords: Auditory feedback; Chronic Obstructive Pulmonary Diseases; Digital Health Technology; Exercise; Exercise adherence; Pulmonary rehabilitation; Mobile applications
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music Walking Application BeatClearWalker (BCW) (Experimental): As it is a single-arm feasibility study, all participants will be allocated to one arm, receiving routine personalised walking exercise while listening to music from the smartphone using the music walking application BeatClearWalker during their Pulmonary rehabilitation Programme.
  Interventions: Device: Music walking application BeatClearWalker (BCW)

INTERVENTIONS:
Device: Music walking application BeatClearWalker (BCW) — The music walking application (BCW) is a smartphone application that can monitor the walking pace and allow individuals to listen to music and give immediate feedback so they can correct their walking pace to match their target walking speed, as prescribed by the healthcare professional. The application provides real-time audio feedback in the form of music; the music sound quality will reduce whenever the walking speed drops below or exceeds the participant's target walking speed. Simply, the application will work to supervise service users while exercising walking. The investigators are trying to assess the feasibility of this application with service users during their Pulmonary Rehabilitation programme (at the hospital/ home) to find out how participants interact with listening to music while exercise walking and how well they're able to keep to their target speed.

SUMMARY:
Pulmonary Rehabilitation (PR) is an evidence-based intervention to effectively manage the physiological and psychological effects of Chronic Obstructive Pulmonary Disease (COPD). The aims of PR are to improve symptoms of COPD, increase exercise capacity, increase independency, improve overall behaviour related to health (like exercising more), and enhance quality of life. The cornerstone of PR programmes is aerobic exercise prescription. Typically, walking exercise is used, and the prescription is individualised for each patient based on their maximal walking exercise capacity. However, adherence to walking exercise is challenging for service users, particularly when unsupervised at home. The use of music during exercise shows promise as a tool to decrease the perception of fatigue and increase motivation, but the integration of music via smartphone applications to support walking exercise adherence during PR has not been explored. This project aims to assess if a new mobile application BeatClearWalker (BCW) intervention is practical, acceptable, and effectively used by people living with COPD. The app is designed to help people living with COPD attending PR adhere to their prescribed walking pace during exercise. The BCW app provides real-time, personalised music feedback through music degradation to optimise the dose of walking exercise.

DETAILED DESCRIPTION:
Previous research has shown that adherence to the prescribed walking exercise intensity is challenging for individuals with COPD and that methods to provide further support are needed. Using activity monitors and trackers to give feedback can increase the walking exercise participation of people living with COPD. However, it has been reported that more than half of steps taken during exercise were below the prescribed pace. It is possible to individually prescribe exercise intensity by deriving cadence (steps taken per minute) from the ISWT and ESWT using activity monitor. Furthermore, activity monitors have been used to measure level of adherence to the intensity of the prescribed walking exercise prescriptions in the context of PR and chronic respiratory diseases.

Listening to music in daily life can decrease stress and improve the psychological well-being. Implementing music to enhance exercise performance has been utilised with different populations. Auditory feedback in the form of listening to music is one example where exercising to music can be utilised as distraction from fatigue perception or used as a motivational tool to exercise in a healthy population. Previous studies have investigated the effect of listening to music while exercising at different intensities and music tempos on fatigue perception and have shown a positive effect in decreasing the perception of fatigue. In addition, the effect of choosing the preferred versus non-preferred music genre on repeated sprints showed significant improvement in motivation to exercise and lower perceived exertion rates in the preferred music genre group. Similarly, in COPD, listening to music as distractive auditory stimuli while exercising decreases breathlessness and fatigue symptoms resulting in increased aerobic capacity and HRQOL. In another study, individuals with COPD who listened to music while performing high-intensity exercise, showed a reduction in dyspnoea, which was associated with higher tolerance of high-intensity exercise as measured by endurance time. The findings of a previous study showed that participants who listened to music can perform significantly more exercise compared to participants who listened to grey noise or silence. Paced walking to music with COPD participants showed significant improvement in dyspnoea, exercise tolerance, HRQoL and fatigue. In the context of unsupervised walking exercise among individuals living with COPD, paced walking to interval beeps sound as such in metronomes to maintain the walking exercise intensity had been investigated previously. In a prospective observational clinical trial, the effect of home-based PR on exercise capacity and HRQoL using paced walking to metronome was investigated. The results showed improvements in maximal exercise capacity (six minute walk test: 6MWT) and HRQoL (SGRQ). However, the constant rhythm such as in metronome style feedback may not be interesting overtime which can make walking exercises less engaging and lead to reduced motivation for long-term adherence.

Combining the effect of paced walking when listening to 'metronome style' feedback and preferred music to support walking exercise might offer a more enjoyable way to coach people living with COPD to walk for exercise at their prescribed intensity. This principle has been investigated in adult without reported diseases population using a mobile application (app), the BeatClearWalker (BCW), as shown in the link (https://youtu.be/MLy4GA8_eUc?si=oQL3mklA2bRKbnQl). The BCW is a fitness smartphone application that monitors walking cadence and helps individuals to walk at their individually-prescribed cadence and maintain that cadence. The app is designed to work on smartphones run by Android software only. Despite a considerable number of fitness applications that monitor walking distance, this is the first application designed to support walking and provide real-time feedback about cadence through music sound quality. The application allows service users to listen to any music while walking and apply dynamic live audio feedback to help individuals to walk at and maintain the pre-set individualised target walking cadence which can be entered on the application. The real-time, hands-free audio feedback is noticeable and designed to disrupt the quality of the played music. The feedback comes in two forms: (1) clear music, similar when listening to any typical music played in streaming music player or (2) degradation of music audio quality. The music will play without effect if the individuals walk at or above their targeted cadence. Once the walking cadence drops below the targeted, the quality of the music will be degraded and will return to normal once the individual reaches the targeted cadence again.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent for participation in the study.
* The patient is referred for PR at the UHL.
* The patient has a confirmed diagnosis of COPD using spirometry (based on GOLD criteria)
* Male or female, aged 18+ years.
* Able to communicate in written and spoken English.

Exclusion Criteria:

* Unable to provide valid informed consent.
* Lack of motivation to participate in PR programme.
* Any-contra-indications absolute or relative to exercise training.
* Has had a cardiac event within last 6 weeks
* Severe psychiatric disorders
* Patients with a history of MRSA +ve screens (patients can be assessed and given an exercise programme but cannot attend the classes. Patients need to have 3 consecutive -ve MRSA swabs before they can attend).
* Unable to understand written or spoken English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-09-12 (Estimated); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
The proportion of recruited participants who do not use the BCW app. | Post PR 6-8 weeks.
The proportion of recruited participants who complete the follow-up assessment. | Upon the completion of the PR programme at 6-8 weeks.
The proportion of patients who meet the eligibility criteria. | 11 months
  The percentage of eligible from those who were screened against the eligibility criteria
The proportion of individuals with COPD who express interest in participating in the study. | 11 months
The proportion of eligible participants who provide consent to enrol. | 11 months
  After meeting the eligibility criteria at the screening stage.

SECONDARY OUTCOMES:
Medical Research Council (MRC) Dyspnoea Scale | Baseline (Pre-PR) and Follow-up (Post-PR, at 6-8 weeks).
  Medical Research Council (MRC) Dyspnoea Scale , measuring the level of breathlessness.
  Scale: Minimum value: 1 Maximum value: 5. The higher the score, the worse the outcome (breathlessness).
Generic Health Status Questionnaire (EQ-5D-5L) | Baseline (Pre-PR) and Follow-up (Post-PR, at 6-8 weeks).
  The EQ-5D-5L evaluates generic health status, with five dimensions of health assessed.
  Scale: The descriptive system results in a single score; higher scores generally indicate worse outcomes.
Generalized Anxiety Disorder 2-item (GAD-2) | Baseline (Pre-PR) and Follow-up (Post-PR, at 6-8 weeks).
  The Generalized Anxiety Disorder-2 (GAD-2) is a brief screening tool for generalized anxiety disorder, measuring the frequency of anxiety symptoms over the past two weeks.
  Scale: Minimum score is 0, and Maximum score is 6. Higher scores indicate worse anxiety symptoms.
  A score of 3 points is the preferred cut-off for identifying possible cases and in which further diagnostic evaluation for generalized anxiety disorder is warranted.
Generalized Anxiety Disorder 7-item (GAD-7) | Baseline (Pre-PR) and Follow-up (Post-PR, at 6-8 weeks).
  The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item scale that measures the severity of generalized anxiety disorder symptoms over the past two weeks.
  Scale: The following cut-offs correlate with level of anxiety severity:
  Score 0-4: Minimal Anxiety Score 5-9: Mild Anxiety Score 10-14: Moderate Anxiety Score greater than 15: Severe Anxiety
Walking exercise time at an individually prescribed cadence over the total time spent in walking exercise (Percent). | Data collected after each walking exercise session during the PR programme (6-8 weeks).
  Data of the walking exercise will be collected during PR from BCW exercise log.
Walking exercise time below the individually prescribed cadence. (Percent) | Data collected after each walking exercise session during the PR programme (6-8 weeks).
  Data of the walking exercise will be collected during PR from BCW exercise log.
The proportion of time spent walking over the prescribed walking exercise duration as measured during the Endurance Shuttle Walking test. (Percent) | Data collected after each walking exercise session during the PR programme (6-8 weeks).
  Data will be collected after each walking exercise session during PR from BCW exercise log.
Exercise Adherence Rating Scale (EARS). | Follow-up (Post-PR, at 6-8 weeks).
  It will assess the adherence levels of individuals to their exercise prescription. Scale: The score range, 0 to 24. Higher scores generally indicate better adherence (24 indicates best adherence). The scale will be used post pulmonary rehabilitation programme
Walking exercise time above the prescribed cadence. (Percent) | Data collected after each walking exercise session during the PR programme (6-8 weeks).
  Data of the walking exercise will be collected during PR from BCW exercise log.
Exercise Capacity test (Incremental Shuttle Walking test [ISWT]) | Baseline (Pre-PR) and Follow-up (Post-PR, at 6-8 weeks).
  Incremental Shuttle Walking Test, Distance walked in meters
Exercise Capacity (Endurance Shuttle Walking test [ESWT]) | Baseline (Pre-PR) and Follow-up (Post-PR, at 6-8 weeks).
  Endurance Shuttle Walking Test (ESWT), Time walked in seconds.
Patient Health Questionnaire-9 (PHQ-9) | Baseline (Pre-PR) and Follow-up (Post-PR, at 6-8 weeks).
  The Patient Health Questionnaire-9 (PHQ-9) measures the severity of depression based on 9 criteria over the past 2 weeks.
  Scale: Minimum score: 0, Maximum score: 27. Higher scores indicate more severe depressive symptoms.
  Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
CRQ-SR (Chronic Respiratory Questionnaire - Self-Reported) | Baseline (Pre-PR) and Follow-up (Post-PR, at 6-8 weeks).
  Chronic Respiratory Questionnaire - Self-Reported (CRQ-SR) measures quality of life in individuals with chronic respiratory diseases.
  Scale: Minimum and maximum values vary by subscale. Higher scores indicate better health-related quality of life.
Patient Health Questionnaire-2 (PHQ-2) | Baseline (Pre-PR) and Follow-up (Post-PR, at 6-8 weeks).
  The Patient Health Questionnaire-2 (PHQ-2) measures the frequency of depressed mood and anhedonia over the past 2 weeks.
  Scale: A PHQ-2 score ranges from 0-6. A score of 3 as the optimal cutpoint when using the PHQ-2 to screen for depression. If the score is 3 or greater, major depressive disorder is likely.
COPD Assessment Test (CAT) | Baseline (Pre-PR) and Follow-up (Post-PR, at 6-8 weeks).
  The COPD Assessment Test (CAT) evaluates the impact of COPD on the individual life.
  Scale: Minimum score: 0, Maximum score: 40. Higher scores indicate worse health status.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Orme, PhD, Principal Investigator — University of Leicester; Linzy Houchen-Wolloff, PhD, Study Director — NIHR Leicester Biomedical Research Centre - Respiratory, University Hospitals of Leicester NHS Trust; Sally J Singh, PhD, Study Chair — NIHR Leicester Biomedical Research Centre - Respiratory, University Hospitals of Leicester NHS Trust
Locations (2):
- United Kingdom (2):
  - NIHR Leicester Biomedical Research Centre - Respiratory, Leicester, Leicestershire
  - University Hospitals of Leicester (UHL), Leicester, Leicestershire

IPD SHARING:
Plan to Share IPD: No